CLINICAL TRIAL: NCT05431244
Title: Pilot Study of Antiviral Treatment in Combination With Low-dose Gemcitabine in EBV-associated Gastric Cancer (EBVaGC)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research withdrawal before patient registration due to difficulty in continuing research
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-03-110
Record Dates: First submitted 2022-06-13; First posted 2022-06-24 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Antiviral treatment in combination with low-dose gemcitabine (Other): For 1st & 2nd cycle D1, 8, 15 Gemcitabine 30-300mg/m2 IV over 30 minutes D8-28 Valganciclovir 900mg qd Every 4 weeks
  For 3rd ~ 6th cycle D1, 8, 15 Gemcitabine 30-300mg/m2 IV over 30 minutes D1-28 Valganciclovir 900mg qd Every 4 weeks
  Interventions: Drug: Antiviral treatment in combination with low-dose gemcitabine

INTERVENTIONS:
Drug: Antiviral treatment in combination with low-dose gemcitabine — -maximun 6 cycles Gemcitabine; 30mg/m2 or 100mg/m2 or 300mg/m2 D1,D8, D15 (Q 1 week,3 times, rest for 1 week, every 4 weeks ) 1,2 cycle Valganciclovir; 900mg D8~D28 (from 1 week after Gemcitabine iv started, qd, PO, 21days) 3~6cycle Valganciclovir; 900mg D1~D28 (from Gemcitabine start date, PO, 28days)

SUMMARY:
Epstein-Barr virus (EBV) is a double-stranded DNA human gamma herpes virus that establishes a persistent infection in over 90% of individuals. Most infections are self-limiting, but some cases are associated with the development of malignancies of lymphoid or epithelial origin. EBV-associated gastric carcinomas (EBVaGC) make up about 9% of all stomach cancers.

The constant presence of the viral genome in EBVaGC suggests the applicability of novel EBV-targeted therapies.

The antiviral nucleoside drug, (val)ganciclovir (GCV), is effective only in the context of the viral lytic cycle in the presence of EBV-encoded thymidine kinase (TK)/ protein kinase (PK) expression. JM Lee et al. reported that gemcitabine was lytic inducer via activation of the ATM/p53 genotoxic stress pathway in EBVaGC and confirmed the efficacy of gemcitabine-GCV combination treatment.

So we planned this proof of concept trial to apply the antiviral agent in EBVaGC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥20 years of age.
* Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after second-line therapy.
* The patient's tumor tissue must have the pre-defined characteristics as follows ; EBV+
* ECOG performance status 0-1
* Patients must have a life expectancy ≥ 4 months from proposed first dose date.
* The patient has measureable or evaluable disease as determined by standard computed tomography (CT) or magnetic resonance imaging (MRI) imaging. Examples of evaluable, nonmeasurable disease include gastric, peritoneal, or mesenteric thickening in areas of known disease, or peritoneal nodules that are too small to be considered measurable by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below: WBC ≥ 3,500 cells/mm3 and ≤ 50,000 cells/mm3, ANC ≥ 1,500 cells/mm3, Hemoglobin ≥ 9 g/dL (transfusion allowed), Platelet count ≥ 100,000 /mm3; Total bilirubin ≤ 1.5 X ULN, AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN; Creatinine clearance ≥60 mL/min
* Provision of fully informed consent prior to any study specific procedures.

Exclusion Criteria:

* The patient has a history severe or unstable heart disease, e.g. coronary artery disease requiring increased dose of anti-anginal medication and/or coronary angioplasty (including stent placement) within 24 months ( congestive heart failure NYHA III or IV, unstable angina, history of myocardial infarction within the last 12 months, clinically significant arrhythmia)
* The patient is pregnant or breastfeeding.(For women with pregnancy potential, an effective method of contraception should be agreed.)
* The patient has ongoing Uncontrolled systemic diseases (diabetes, hypertension, hypothyroidism, infection, etc.)
* The patient has ongoing central nervous system malignancy. (except for lesions that have been completely removed or underwent anterior brain radiotherapy/gamma knife procedure)
* The patient has a history of allergic reactions to gemcitabine, Valganciclovir, aciclovir, valacyclovir ganciclovir
* Patients with interstitial pneumonia or pulmonary fibrosis with clinical symptoms

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24months
  Modified RECIST 1.1 criteria will be used to assess patient response to treatment by determining PFS and ORR. The modified RECIST 1.1 guidelines for measurable, non-measurable, target and non-target lesions and the objective tumour response criteria

SECONDARY OUTCOMES:
Best Overall Response Rate (BOR) | up to 24months
  Modified RECIST 1.1 criteria will be used to assess patient response to treatment by determining PFS and ORR. The modified RECIST 1.1 guidelines for measurable, non-measurable, target and non-target lesions and the objective tumour response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, M.D. Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No